CLINICAL TRIAL: NCT05432440
Title: Evaluation of Pharmacist-guided Digital-based Asthma Education for Indonesian Children With Asthma
Acronym: MIRACLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Made Ary Sarasmita, Clinical Pharmacist, Department of Pharmacy, Faculty of Mathematics and Science, Udayana University; PhD student, Department of Clinical Pharmacy, Taipei Medical University, Taipei, Taiwan, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1368/LT/2022
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Asthma in Children; Asthma Chronic; Asthma
Keywords: asthma; children; serious game
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: After informed consent provision and baseline assessment, participants will be allocated into two groups, including the intervention group (IG) and the control group (CG). The intervention will be a computer-based asthma self-management education entitled Module of Inhaler and Asthma Triggers for Children (MIRACLE) and usual care. It will consist of interactive narratives and a serious game, an asthma action plan, and a video of the inhaler technique. The control group will receive a paper-based asthma education (booklet) and usual care. The study duration will be set for 2 months by applying those media for 7 days at home and the minimum required time for using the MIRACLE program will be 15 minutes per day. Two groups will be equipped with a peak flow meter and an asthma action plan, and they will be encouraged to write their daily symptoms and activities in a diary.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors for collecting outcome data at 1 and 2 months will be masked to group allocation. They will also be prohibited to contact patients directly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (the digital asthma education program) (Experimental): The intervention group receives the digital asthma education program (MIRACLE program). It consists of an asthma interactive narrative, a serious game, and an asthma action plan. It mainly covers asthma self-management and asthma attack prevention, such as asthma definition, asthma triggers and how to prevent asthma triggers exposures, asthma medications, proper inhaler technique, and asthma written action plan.
  The time schedule will be described as:
  1. Explain study purposes, program, procedures, and instructions (10 minutes).
  2. Accompany children and parents to download and install the MIRACLE program on Google Play Store for free on their personal computers, tablets, or smartphones (5 minutes).
  3. Asthma education will take place over one session lasting approximately 45 minutes.
  Interventions: Behavioral: The digital asthma education program
- Control group (the booklet asthma education program) (Active Comparator): For the control group, a pharmacist (same personnel) will provide an asthma education using a booklet for 45-60 minutes to children and parents. Patients will be asked to read the booklet at home for 15 minutes in 7 days. It mainly covered the same content as the MIRACLE program. The time schedule will be described as:
  1. Explain study purposes, booklet, procedures, and instructions (10 minutes).
  2. Asthma education will take place over one session lasting approximately 45 minutes.
  Interventions: Behavioral: The digital asthma education program

INTERVENTIONS:
Behavioral: The digital asthma education program — The intervention group receives the digital asthma education program (MIRACLE program). It consists of an asthma interactive narrative, a serious game, and an asthma action plan. It mainly covers asthma self-management and asthma attack prevention, such as asthma definition, asthma triggers and how to prevent asthma triggers exposures, asthma medications, proper inhaler technique, and asthma written action plan.

SUMMARY:
Poor adherence and self-management in children with asthma results in poorly controlled asthma and increased morbidity. Pharmacists could take important roles in delivering asthma education to ensure that children can manage their disease. This study aims to evaluate the effectiveness of improving asthma control, knowledge, and quality of life. An open, randomized controlled trial will be conducted to evaluate the effectiveness of pharmacist-led digital-based asthma self-management education for children with asthma compared with paper-based asthma self-management education. Recruitment of the participants will be held at the outpatient ward of the Department of Paediatrics in 4 public hospitals in Bali Province, Indonesia, including Sanglah Public Hospital, Denpasar City; Wangaya Public Hospital, Denpasar City; Mangusada Public Hospital, Badung Regency; and Udayana University Hospital, Badung Regency. Participants will be provided with informed consent, then randomly divided into either a control group or an intervention group.

The following will be the hypotheses of the study:

1. The intervention group receiving the MIRACLE education program has a better asthma control compared to the control group.
2. The intervention group receiving the MIRACLE education program has a greater improvement in asthma quality of life compared to the control group.
3. The intervention group receiving the MIRACLE education program has a better understanding of asthma knowledge in general compared to the control group.
4. The intervention group receiving the MIRACLE education program has a better performance in practicing inhaler techniques compared to the control group.
5. The intervention group receiving the MIRACLE education program has fewer unscheduled visits to the hospital and less hospitalization compared to the control group.
6. The intervention group receiving the MIRACLE education program will be satisfied with the digital asthma education.

DETAILED DESCRIPTION:
Description A randomized controlled trial will be conducted in four teaching hospitals in Bali, Indonesia. The module on inhalers and asthma triggers (MIRACLE) had been developed using cultural adaptation and growth mindset elements for Indonesian children with asthma. It consists of an interactive narrative and a serious game. The intervention group will receive the MIRACLE program and written asthma plan, and the control group will receive an asthma booklet. A pharmacist will deliver the education to both groups.

Randomization and Allocation Recruited participants will be allocated to the intervention or control group on a 1:1 basis. Randomization and allocation will be conducted at each research site. Assignment numbers will be printed and sealed in opaque envelopes according to a predefined order. The envelopes will be stored in a secured cabinet. Block randomization will be performed on the basis of 2 units and random numbers will be generated using a random allocation software program by an external researcher not involved in the study. The block size will be confidential. Group assignment will be concealed until children and parents complete the consent procedures. At the time of recruitment, the researchers coordinating this study will open the numbered envelope and will allocate each participant to the control group (paper-based asthma health education) or the intervention (computer-based asthma education/the MIRACLE program) using a secured computer file. A pharmacist will administer the intervention and will be aware of the allocated groups. Due to the nature of the study, participants may be aware of the existence of the alternative group. To minimize bias, the assessors who will assess the baseline and follow-up measures will not be aware of the allocation.

Sample size calculation We will use G-Power software (version 3.1, Heinrich-Heine-Universität Düsseldorf, Germany) to calculate the estimated sample size of this study. Assuming a power of 80% with a two-sided alpha level of 0.05 to detect the difference between the intervention group and the control group, at least 36 participants were needed for each group. We will anticipate a low rate of follow-up attrition (20% dropout) and consider a sample size of 50 per group, an estimated 100 participants in total.

Study procedures Before study Before conducting the study, one pharmacist will undergo training provided by a certified asthma educator. This study will evaluate a digital-based intervention involving pharmacists in delivering patient education and counseling. A checklist form will be filled out when the pharmacist delivers asthma education to both groups.

Recruitment The recruitment process will be accompanied by pediatricians and nurses in the hospitals. Potentially eligible participants will be identified through 2 pathways: 1) first, the pediatricians will identify all children with asthma visiting the outpatient hospitals on the date of each patient's clinic visit. A research assistant will approach potential participants and will perform screening on the eligibility, then we will provide an explanatory statement, an informed consent, and a child assent form to the patients and parents. Potential participants will be asked to leave their contact details to allow one of the research assistants to contact them, or 2) second, through the electronic medical record (EMR) system in the hospitals, and then identified patients will receive a phone call, a short message, or an email. Written informed consent and child assent form from the patient and parents/guardians will be sought after the explanation procedure. Participation in this study will be voluntary and without any force to them. The subjects have the right to withdraw from the study at any time and there will be no adverse effect on their medical treatments. The reasons for not participating in patients deem ineligible or decline to participate during the follow-up session will be recorded.

Baseline visit (Time 0)

A research assistant will call all patients in advance of their clinic appointment to introduce or reintroduce the study so that they will have enough time to complete the baseline assessment, which lasts approximately 10-15 minutes. Each child will be weighed and measured as part of the polyclinic routine, then will be interviewed by the researcher as they will wait to see the pediatrician. During the assessment, the researchers will be available to answer questions and assist younger children with reading if necessary. The researchers will collect baseline measurements, including:

1. Demographic characteristics, parental information, and disease-related information. At baseline, each child's parents provide demographic details and the information about their child's asthma
2. Asthma control will be measured using Asthma Control Questionnaire (ACQ).
3. Asthma quality of life will be measured using the Paediatric Asthma Quality of Life Questionnaire (PAQLQ).
4. Inhaler techniques will be measured using the Indonesian Counseling for Pharmacy Practice guideline: the inhaler technique checklist.
5. Self-reported expressions of children and parents when dealing with a previous asthma attack.
6. The number of unscheduled visits to the hospital and number of hospitalization for the previous 6 months.
7. Forced expiratory volume in the first second (FEV1) will be measured using a spirometer and a peak flow meter, respectively, according to Indonesian guidelines.
8. Asthma knowledge will be measured by questions provided by the researchers.

Intervention group A pharmacist will provide an asthma education (the MIRACLE program) for 45-60 minutes to children and parents. After face-to-face education, the pharmacist will ask patients to read the narrative and play the game. This activity will be continued at home for 7 days, and 15 minutes per day will be a minimal requirement. It mainly covers asthma self-management and asthma attack prevention, such as asthma definition, asthma triggers and how to prevent asthma triggers exposures, asthma medications, proper inhaler technique, and asthma written action plan. For the control group, a pharmacist (same personnel) will provide an asthma education using a booklet for 45-60 minutes to children and parents. Patients will be asked to read the booklet at home for 15 minutes in 7 days. It mainly covered the same content as the MIRACLE program.

Follow-up (Time 1 and Time 2) Outcome measures will be collected at the baseline and at 1 and 2 months (T1 and T2) from the baseline to allow comparisons. Identical data collection forms will be used for both groups. The outcome assessors for collecting outcome data at 1 and 2 months will be masked to group allocation. They will also be prohibited to contact patients because any interaction might lead to study bias. Data collection will be ended as all participants completely finished the 2-month measurement period. One month and two months after the intervention, all of the children in the study will be visited at home, and baseline measures will be repeated (ACQ, PAQLQ, FEV1, knowledge, correct inhaler techniques, asthma experiences). Children will be asked to express their satisfaction with the digital tools. Parents will be asked to rate their child's unscheduled visits, and admissions to the hospital, and they will be asked to share their experiences with asthma.

Analysis Descriptive analysis will be undertaken to analyze the demographic characteristics as appropriate in both groups. Any difference in baseline characteristics between groups will be accounted for in the statistical analysis. The baseline characteristics of the two groups will be compared using the student's t-test for normally distributed continuous variables (mean, SD), or Mann-Whitney U test for non-normally distributed continuous variables (median, interquartile range [IQR]), and chi-square or Fischer's exact test for categorical variables (percentages). A chi-square test will be used to analyze sex, age, level of mother education, and history of asthma to determine whether significant differences existed between the two groups.

The study follows intention-to-treat analysis and a common threshold two-sided p-value (P<0.05) for statistical significance interpretation. In addition, Cohen's d for determining effect size will be calculated. Cohen's d is an effect size to indicate a standardized difference between two means with the interpretation of Cohen's d of >0.8, >0.5, and <0.2 indicating large effect, moderate effect, and poor effect, respectively. Asthma control and asthma quality of life scores at the baseline and follow-up will be compared by paired samples t-test. Correct inhaler technique before and after the intervention will be compared with Pearson's Chi-square test. We will compare the outcomes before and after the study using paired t-tests for the continuous variables and the McNemar test for the dichotomous outcomes variables. We will use Wilcoxon signed-rank tests for comparisons of nonparametric paired continuous data. Mann-Whitney tests will be used for univariate comparisons between groups for the number of emergency visits, the number of hospitalization, and the number of school absences. Statistical analysis will be performed using SPSS software (version 23.0; SPSS Inc., Chicago, IL, USA).

Missing data and dropouts Patients will be rated as dropouts when they are excluded from the study at their own request or if they are no longer able to participate in the study until the final visit. Patients who are not able to undergo all measurements during the follow-up visits will remain in the study. Multiple imputation methods will be used to impute missing data with less than 25% missing values. This is typically more efficient than a complete case analysis when covariates have missing values.

ELIGIBILITY:
Inclusion Criteria:

1. Children with asthma, asthma was diagnosed by a medical doctor, pediatrician, or medical records.
2. Children with asthma in the range age of 6 - 13 years old.
3. Had a history of asthma or had a previous asthma attack in 1 year.
4. Able to communicate in Bahasa Indonesia and pose to use a computer, tablet, or smartphone.
5. No serious cognitive impairments.
6. Agree to participate in the study and follow the instructions.

Exclusion Criteria:

1. Disagree to participate in the study.
2. Had another history of respiratory diseases or conditions that may affect responses.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Control as assessed by Asthma Control Questionnaire (ACQ). | 2 months
  The primary outcome will be the changes in asthma control. The Indonesian version of the Asthma Control Questionnaire (ACQ, proposed by Juniper et al, 1995) is a validated measure of a patient's abilities to control asthma. It composes of 5 questions about asthma symptoms, 1 question about bronchodilator use during the previous week, and 1 question about FEV1% change. All questions will be scored 0 to 6, and a total score will be expressed as the mean of these scores. Asthma control will deteriorate as the score increase. A clinically important change in ACQ score will be reported to be 0.5. If the post-test score will be lower than the pretest score, it will be indicated that asthma control will be improved. Patients will be asked to recall their experiences during the previous 7 days and will respond to the questions using a 7-point scale.

SECONDARY OUTCOMES:
Asthma Quality of Life assessed by Pediatric Asthma Quality of Life Questionnaire (PAQLQ) | 2 months
  Asthma quality of life will be measured using validated the Indonesian version of the Pediatric Asthma Quality of Life Questionnaire (PAQLQ). It consists of 23 questions covering symptoms, activities, and emotions related to asthma. Each item will be scored on a 7-point scale and will be averaged for a total mean score, with higher scores indicating a better asthma-related quality of life. When administering the questionnaire, it is important to explain to children that the PAQLQ will measure the problems that many children with asthma find troublesome. The best score is 7.0, which interprets as the patient has no impairments due to their asthma.
The level of asthma knowledge, assessed by Asthma Knowledge Questions | 2 months
  Asthma knowledge questions were developed by the experts panel while developing the content of asthma education. It includes 20 true/false questions covering asthma triggers, asthma symptoms, asthma treatment, and asthma management. Total possible scores ranged from 0 to 20, with higher scores indicating greater asthma knowledge. It will be considered to be knowledgeable (75% of the correct answers), quite knowledgeable (50% the correct answers), less knowledgeable (<50% the correct answers).
Number of Correct Inhaler Techniques Performance, assessed by Indonesian Inhaler Practice Checklist | 2 months
  participants will be asked to demonstrate how they actually use their device. For this purpose, a placebo in the form of a metered-dose inhaler (MDI) device will be used. Correctness of inhaler use will be assessed using pre-defined checklists based on the Indonesian Counseling and Pharmacy Practice Guideline: Inhaler Practice Checklist (2008). The correct inhaler technique will be defined as the correct performance of every step on the checklist. Incorrect inhaler use will be defined as the 1 or more steps done incorrectly. A total score will be calculated with 0 (incorrect application) and 1 (correct application). Possible errors will be corrected by verbal instructions and a visual demonstration. For ethical reasons, the correction will be performed in both groups. Children will demonstrate their inhalation technique until it will be performed correctly.
number of unscheduled visits | 2 months
  number of unscheduled visits to the hospital or emergency department due to asthma exacerbation
number of hospitalization | 2 months
  number of hospital admission during the study due to asthma exacerbation. a number of hospitalization will be reported descriptively.
number of school absences | 2 months
  number of school absences due to asthma exacerbation. The number of school absences will be reported descriptively.
self-reported medication adherence, assessed by self-reported medication adherence checklist | 2 months
  Medication adherence will be recorded using the number of prescriptions refilled. Respondents indicate how often they engage in the four non-adherent behaviors on a 1-to-5 frequency scale (always, often, sometimes, rarely, or never), with higher scores relating to better adherence. The result will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang Yi Chen, Prof, Study Chair — Taipei Medical University
Locations (4):
- Indonesia (4):
  - Mangusada Teaching Hospital, Badung, Bali
  - Udayana University Hospital, Badung, Bali
  - Sanglah General Hospital, Denpasar, Bali
  - Wangaya Teaching Hospital, Denpasar, Bali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarasmita MA, Larasanty LPF, Kuo LN, Cheng KJ, Chen HY. A Computer-Based Interactive Narrative and a Serious Game for Children With Asthma: Development and Content Validity Analysis. J Med Internet Res. 2021 Sep 13;23(9):e28796. doi: 10.2196/28796. PMID 34515641